CLINICAL TRIAL: NCT02987686
Title: Topical Infliximab for the Treatment of Sterile Corneal Melt
Brief Title: Topical Infliximab for Sterile Corneal Melt
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de recherche en ophtalmologie de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE16.221
Record Dates: First submitted 2016-10-26; First posted 2016-12-09 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Sterile Corneal Melt
Keywords: Topical Infliximab; Cornea; Keratolysis
MeSH Terms: conditions — Corneal Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Infliximab (Experimental): Additionally to standard treatment, patients with all inclusive criteria and none exclusive criteria will be included in the therapeutic group and will receive topical infliximab QID for 4 weeks.
  Interventions: Drug: Topical Infliximab
- Observational group (No Intervention): Patients with all inclusive criteria and one exclusive criteria will receive the standard treatment, without topical infliximab.

INTERVENTIONS:
Drug: Topical Infliximab — Aside from the standard treatment, patients will receive topical infliximab ( 10mg/ml) four (4) time per day for four (4) weeks.
  Other Names: Remicade
  Arms: Topical Infliximab

SUMMARY:
Corneal melt is a complication that could affect very ill eyes and lead to the thinning of the cornea (the clear window covering of the eyes). This thinning can lead to severe consequences such as the leakage of the liquid inside the eye (ocular perforation), or even blindness. Corneal melt can be caused by certain infections or as a sterile process. This project only includes patients with a sterile corneal melt (without an infection) caused by diseases such as rosacea, Sjogren's syndrome, rheumatoid arthritis, Crohn's disease, Stevens Johnson syndrome, as well as toxic epidermal necrolysis or mucous membrane pemphigoid.

Infliximab is an antibody against tumour necrosis factor alpha and has been used to treat or prevent corneal melt in certain patients with inflammatory of auto-immune disease. In this situation, infliximab was used intravenous (using veins) in order to treat the whole body.

This study's hypothesis is that infliximab can safely be used as eye drops for the treatment of sterile corneal melt.

DETAILED DESCRIPTION:
This is an unmasked, prospective, single-center trial of twelve patients with sterile corneal melt and an underlying auto-immune or inflammatory disease, such as rosacea, Sjogren's syndrome, rheumatoid arthritis, Crohn's disease, Stevens Johnson syndrome, as well as toxic epidermal necrolysis or mucous membrane pemphigoid.

The aim of this phase I study is to evaluate the safety and tolerability of topical infliximab 10mg/ml eye drops for the treatment of corneal melt. As such, six (6) subjects will be recruited in the experimental treatment study and six (6) subjects will be enrolled in the parallel observational study. Indeed, candidates having all inclusion criteria but one exclusion criteria (which are contraindication to infliximab use), will be recruited in the observational study, will receive the standard treatment without infliximab.

During the treatment period, subjects in the therapeutic study will receive topical infliximab 10mg/ml four (4) times per day for four (4) weeks. In order to determine the safety profile, potential side effects as well as the course of the disease, subjects will be monitored while on the study medication as well as for 8 weeks following discontinuation of the drug. The ophthalmological follow-up will be identical in the two groups. However, only subjects enrolled in the experimental treatment study will receive additional laboratory tests. The total study duration for each patient will be 12 weeks.

In terms of statistical analysis, the investigators will focus on describing the outcome measured in the study. For instance, the investigators will describe the number and proportion of side effects, the number of patients with a quiescent corneal melt at 4 weeks and the patients who required a tectonic surgery at 12 weeks post-treatment. The investigators will report the average and standard of deviation of the OSDI score, the epithelial deficit surface as well as the minimal corneal thickness. Moreover, the investigators will perform exploratory statistical analysis in order to study the disease course of each subject and comparing the addition of infliximab to the standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years;
* Any degree of active sterile corneal melting , as documented by slit-lamp examination, showing an epithelial defect and stromal thinning;
* Negative work-up for local and systemic infectious causes
* Negative corneal cultures (may show growth of common contaminants)
* Capable of providing informed consent;
* Capable of administering eye drops either themselves or through a caregiver.

Exclusion Criteria:

* Any active ocular or systemic infection including active or latent tuberculosis, histoplasmosis, coccidiomycosis, cytomegalovirus, pneumocystosis, aspergillosis, or hepatitis B.
* History of neoplasia diagnosed within the last 5 years
* Demyelinating disease
* Diabetes
* Congestive heart failure
* Significant anomalies on complete blood count, creatinine or hepatic enzymes
* Pregnancy or breast feeding
* Allergy to infliximab or to the drug vehicle (Refresh liquigel)
* Past or present use of anti-TNF-α medications or human interleukin-1 receptor antagonist (anakinra, IL-1Ra)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 weeks
  Number and type of adverse events
Percentage of patients finishing 4 weeks of infliximab use | 4 weeks
  Percentage of patients finishing 4 weeks of infliximab use

SECONDARY OUTCOMES:
Visual Acuity | 4 and 12 weeks
  Visual Acuity is measured using a Snellen chart
Ocular surface symptoms as assessed by ocular disease index score | 4 and 12 weeks
  Ocular surface symptoms as assessed by ocular disease index score
Conjunctival hyperemia using a slit-lamp photographs | 4 and 12 weeks
  Conjunctival hyperemia using a slit-lamp photographs
Corneal thickness as measured by anterior segment optical coherence tomography | 4 weeks
  Corneal thickness as measured by anterior segment optical coherence tomography
Surface area of the corneal melt using a slit-lamp photographs | 4 weeks
  Surface area of the corneal melt using a slit-lamp photographs
Quiescent corneal state | 4 weeks
  Percentage of eyes presenting a quiescent corneal state at 4 weeks
Eyes requiring tectonic surgery | 12 weeks
  Percentage of eyes requiring tectonic surgery at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Robert, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No